CLINICAL TRIAL: NCT05066347
Title: REmote Cardiac MOnitoring of At-risk SYNCope Patients After Emergency Department Discharge - A Multicenter Randomized Controlled Trial: REMOSYNCED
Brief Title: REmote Cardiac MOnitoring of At-risk SYNCope Patients After Emergency Department Discharge -RCT
Acronym: REMOSYNCED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3781
Record Dates: First submitted 2021-09-21; First posted 2021-10-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Syncope
Keywords: Syncope; Cardiac monitoring; Emergency Department
MeSH Terms: conditions — Syncope; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients randomized to usual care will receive all care as prescribed by the discharging physician and there will be no study specific interventions. The current usual care varies from no outpatient monitoring to short-term Holter monitoring (24 hours to 72 hours).
- Prolonged 24/7 live outpatient cardiac rhythm monitoring (Experimental): Patients randomized to the intervention arm will receive 24/7 live cardiac rhythm monitoring for 15 days. If a patient is randomized to the intervention arm and was prescribed outpatient cardiac monitoring such as Holter monitor, this will be replaced by the 24/7 live monitoring and will be applied either prior or within 24 hours of discharge from the ED.
  Interventions: Device: Cardiophone Plus

INTERVENTIONS:
Device: Cardiophone Plus — Cardiophone Plus (Bittium Faros 360 Mobile event recorder, Bittium Biosignals Ltd., Finland., an external loop recorder with 3 leads for 2 channels. Cardiophone Plus evaluates all cardiac beats and rhythm abnormalities that are detected as per the algorithm programmed into the device. These abnormalities are then automatically and immediately transmitted to a central monitoring station without the need for any patient intervention (device-triggered transmission). This transmission occurs through the cell phone that comes with the device. The central monitoring station is in Windsor, Ontario (Canadian Cardiac Care) and is staffed round the clock by certified electrocardiographic technicians and a cardiologist on-call.
  Arms: Prolonged 24/7 live outpatient cardiac rhythm monitoring

SUMMARY:
Syncope (fainting) is a common reason for emergency department (ED) presentation. Fainting can be caused by heart conditions such as irregular heart rhythm (arrhythmia) that can be life-threatening, structural heart problems, or serious conditions not related to the heart. The standard or usual treatment for the majority of patients at-risk for irregular heart rhythm is getting discharged home with no heart rhythm monitoring. If patients receive any monitoring, only Holter monitoring device that records all heart beats for 24 hours to 72 hours will be used. One-third to half of irregular heart rhythm will be identified only after patients are either discharged from the ED or hospitalized in an inpatient unit. One-third to half of irregular heart rhythm will be identified only after patients are either discharged from the ED or hospitalized in an inpatient unit. The study hypothesize that prolonged live cardiac rhythm monitoring (15 days) of at-risk syncope patients, discharged from the ED, will lead to identification of irregular heart rhythm, which can lead to improved patient safety and lower healthcare costs.

DETAILED DESCRIPTION:
Syncope is defined as a sudden, transient loss of consciousness followed by spontaneous complete recovery.14 It is caused by transient global cerebral hypoperfusion due to decreased cardiac output, excessive vasodilatation, or both. The most common causes include a)reflex (i.e., vasovagal syncope); b)cardiac syncope; and c)orthostatic hypotension. Syncope accounts for 1-3% of ED visits and ~6% of admissions from the ED to the hospital. Each year, syncope accounts for approximately 160,000 ED visits in Canada, with direct hospital costs of approximately $130 million.

ED management of syncope: Overall, up to 10% of patients seen in the ED for syncope will have serious underlying conditions e.g., serious arrhythmia, myocardial infarction, significant hemorrhage, pulmonary embolism] identified and/or die from these conditions within the next 30 days. Until recently, valid and reliable evidence to inform these decisions has been lacking. Professional medical societies in Europe and North America have long called for the development of practical and accurate tools to stratify patients into low, intermediate, and high-risk groups to aid in management decisions. One-third to half of these serious conditions will be identified ONLY AFTER they are either discharged from the ED or hospitalized in an inpatient unit, emphasizing the challenge in risk stratification and ED disposition decision-making. Of these serious conditions that are identified after ED disposition, 68.8% are arrhythmias. While the non-arrhythmias are identified in the first few days after the ED visit, arrhythmias tend to be identified up to two weeks after the ED visit. The hypothesis is that prolonged live cardiac rhythm monitoring of at-risk ED syncope patients, defined as those with CSRS score ≥3 discharged from the ED, will lead to the identification of important arrhythmia or ruling out an arrhythmic etiology and consequently to improved patient safety and lower healthcare costs.

Preliminary work: Two large multicentre prospective studies were completed to derive and validate the Canadian Syncope Risk Score (CSRS) by enrolling 8176 patients from 11 Canadian EDs in whom no serious condition was identified during the index ED evaluation. The CSRS was developed conforming to both methodological standards for clinical decision tool development and reported as per the Transparent Reporting of a Multivariable Prediction Model for Individual Prognosis or Diagnosis (TRIPOD) guideline. Overall, 9.0% of patients were hospitalized and 3.6% suffered 30-day serious outcomes after ED disposition. The CSRS score ranges from -3 to +11. The risk categories were simplified into low, medium, and high, and the 30-day serious outcomes for each of the three risk categories. The incidence of arrhythmias in the medium and high-risk groups were 4.9% and 18.0% respectively. Given the importance of occult arrhythmia and uncertainty regarding the optimal duration of cardiac monitoring, the time interval was analyzed from ED arrival to arrhythmia detection/intervention or unexplained death, and found that half of all arrhythmic outcomes were identified within 2 hours among low-risk patients and within 6 hours among medium- and high-risk patients. Furthermore, the more serious, ventricular arrhythmias occurred only in medium and high-risk patients, and 92% of all arrhythmias among these risk groups were identified within 15 days. These latencies are highly relevant to decisions regarding the utility of cardiac monitoring during and after an ED visit for syncope, with implications for the rational deployment of emerging technology such as outpatient telemetry which permits real-time identification of serious arrhythmias. The above inferences regarding cardiac rhythm monitoring are based on the secondary analysis of observational data. There are no previous randomized controlled trials (RCTs) that assess the role of outpatient prolonged cardiac monitoring to detect occult arrhythmias among CSRS medium and high-risk syncope patients discharged from the ED.

There is a wide variations in ED management, including admission rates (ranging from 5.3% to 19.6% among sites) and outpatient cardiac testing, very low yield for advanced neuroimaging, and inefficiencies in hospital admission (among those hospitalized, 46.5% were for suspected arrhythmias, of whom 71.2% had no cause for syncope identified during hospitalization. Analyzing our cohort, the study found that CSRS low-risk patients will benefit the least from hospitalization and CSRS high-risk patients the most. Currently, 21.6% of CSRS medium-risk patients are hospitalized primarily because of concern for underlying arrhythmia, yet the mortality and the likelihood of identifying an underlying ventricular arrhythmia within 30 days among these patients is very low. Advances in ambulatory cardiac rhythm monitoring suggest that this group is an ideal target for outpatient monitoring, forgoing hospital. admission after ED assessment. A pilot study was recently with 15-day out-of-hospital live cardiac rhythm monitoring of 72 CSRS medium and high-risk patients and found that live cardiac monitoring of at-risk ED syncope patients is feasible, safe, and acceptable.

Hypothesis: the study hypothesizes that a strategy of prolonged outpatient cardiac rhythm monitoring compared to usual care of at-risk syncope patients, defined as those with CSRS score ≥3 when discharged from the ED will lead to improved detection of arrhythmias that require treatment and improve patient safety, healthcare efficiency and patient satisfaction. What are the principal research questions to be addressed? The overall objective of this study is to evaluate a strategy of 15-day live cardiac rhythm monitoring versus usual care to improve the identification of an arrhythmia that required treatment among at-risk syncope patients discharged from the ED through a patient-level RCT.

The overall objective of this study is to evaluate a strategy of 15-day live cardiac rhythm monitoring versus usual care to improve the identification of an arrhythmia that required treatment among at-risk syncope patients discharged from the ED through a patient-level RCT.

Trial Design: prospective patient-level multi-center RCT involving 13 participating EDs across Canada. During the trial period, syncope patients will be block randomized to usual care or prolonged outpatient cardiac rhythm monitoring in blocks of variable sizes and stratified by risk scores (3-5, ≥6) and study site.

Patients randomized to usual care will receive all care as prescribed by the discharging physician and there will be no study-specific interventions. Patients randomized to the intervention arm will receive 24/7 live cardiac rhythm monitoring for 15 days (Cardiophone Plus; an external loop recorder). If a patient is randomized to the intervention arm and is prescribed outpatient cardiac monitoring such as Holter monitor, this will be replaced by the 24/7 live monitoring and will be applied either prior or within 24 hours of discharge from the ED. As the intervention arm provides 24/7 live cardiac monitoring which is a higher level of care than the control arm, there is no safety risk to the patients in the intervention arm. Cardiophone Plus evaluates all cardiac beats and rhythm abnormalities that are detected as per the algorithm programmed into the device. These abnormalities are then automatically and immediately transmitted to a central monitoring station without the need of any patient intervention (device-triggered transmission). The central monitoring station is in Windsor, Ontario (Canadian Cardiac Care) and is staffed round the clock by certified electrocardiographic technicians and a cardiologist on-call.

Timeline and follow-up: the study timeline is 18 months of patient enrollment and data collection. The duration of the treatment period for patients in the intervention arm will receive 15 days of cardiac monitoring. All study patients will be followed at Day 30 either by telephone or email and at 1-year through data linkage with the provincial health database.

Embedded observational study: validation of the CSRS ultra-low-risk criteria and to evaluate if the CSRS can be updated to improve its accuracy, ED physician to obtain verbal consent from patients who are lower risk (score <3) for 30-day follow-up and addition of cardiac biomarker using the left-over blood at study centers that are able to accomplish such additional testing for research purposes. These patients will not be enrolled in the randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥ 18 years old) who present with syncope to any of the study EDs (within 24 hours), are classified as medium (3-5,) or high-risk (≥6) as per the CSRS and are being discharged from the ED either by the ED team or the consulting team if consulted to another service. Patients will be enrolled after written consent.
* For the secondary objectives related to the embedded observational study, validation of the CSRS ultra-low-risk criteria and to evaluate if the CSRS can be updated to improve its accuracy, ED physicians will obtain verbal consent from patients who are lower risk (score <3). These patients will not be enrolled in the randomized controlled trial.

Exclusion Criteria:

* Prolonged loss of consciousness (i.e., > 5 minutes),
* Glasgow Coma Scale < 15 in patients without dementia (or a change in the mental status from baseline in those with dementia);
* Witnessed obvious seizure, or head trauma preceding the loss of consciousness; and those who are unable to provide proper details (e.g., alcohol intoxication or other substance use).
* Patients who are hospitalized on their index ED visit and who had an obvious underlying serious condition for the syncope identified during the index ED visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with arrhythmia that required treatment | within 15-days of the index ED visit
  Identification of an arrhythmia that required treatment among at-risk syncope patients discharged from the ED among patients with CSRS score ≥3.

SECONDARY OUTCOMES:
Number of participants with arrhythmias that did not require treatment | within 15-days of the index ED visit; between 16 and 30 days of disposition
  Arrhythmias that did not require treatment
Rate of Mortality | 1-year
  Distinguishing between deaths secondary to another serious condition and due to an unknown cause
Number of participants with non-arrhythmic serious conditions | within 30-days of disposition
  non-arrhythmic serious conditions
Number of return ED visits | 1-year
  Proportion of patients had return ED visits
Rate of Hospitalizations | 1-year
  Proportion of patients hospitalized
Device Insertion | 1-year
  Proportion of patients with device insertions [pacemaker, implantable cardiac defibrillator (ICD), or a combined pacemaker-ICD device]
Any serious outcome | within 30 days
  The occurrence and identification of any serious outcome for lower-risk patients (CSRS score <3).

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Thiruganasambandamoorthy, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - Civic and General Campuses, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No